CLINICAL TRIAL: NCT02140346
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Inhaled RV1729 in Patients With COPD
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Repeat Doses of RV1729 for 28 Days in Patients With COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respivert Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STN002; 2014-000089-23 (EudraCT Number)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 6-(2-((4-amino-3-(3-hydroxyphenyl)-1H-pyrazolo(3,4-d)pyrimidin-1-yl)methyl)-3-(2-chlorobenzyl)-4-oxo-3,4-dihydroquinazolin-5-yl)-N,N-bis(2-methoxyethyl)hex-5-ynamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 28 day repeat dose (low dose) (Experimental)
  Interventions: Drug: RV1729 28 day repeat dose; Drug: RV1729 matching placebo 28 day repeat dose
- 28 day repeat dose (high dose) (Experimental)
  Interventions: Drug: RV1729 28 day repeat dose; Drug: RV1729 matching placebo 28 day repeat dose

INTERVENTIONS:
Drug: RV1729 28 day repeat dose — Safety and tolerability of repeat doses
Drug: RV1729 matching placebo 28 day repeat dose — Safety and tolerability of repeat doses

SUMMARY:
RV1729 is a new medicine being developed for the potential treatment of asthma and smoking related lung disease (also known as chronic obstructive pulmonary disease - COPD). The objective of this study is to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics repeat doses of RV1729 in patients with COPD for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Be a man or a woman of non-child-bearing potential aged 40 to 75 years
* Women of non-childbearing potential must be either amenorrhoeic >1 year with an appropriate clinical profile or permanently sterilised
* Women must agree not to donate eggs (ova, oocytes) from Screening until at least 6 months after the final dose of study medication
* Men must be willing to use one form of contraception (with documented failure rate less than 1%) and agree not to donate sperm from Screening to 90 days post last dose of study agent
* Chronic obstructive pulmonary disease diagnosis with symptoms compatible with COPD for at least 1 year before Screening.
* Severity of disease: subjects who conform to the current severity classification for Global Initiative for Chronic Obstructive Lung Disease (GOLD, 2014) Grade II/III
* On a background therapy of inhaled steroid with or without the addition of long-acting bronchodilators (either long-acting beta agonists [LABAs] or long-acting muscarinic antagonists [LAMAs]).
* Be able to produce an acceptable induced sputum sample at the Screening visit.
* Capable of complying with all study restrictions and procedures including ability to use the study inhaler correctly.
* A current or previous smoker with a smoking history of ≥10 pack years.
* Have a 12 lead ECG recording consistent with normal cardiac function at the Screening visit and pre-dose Day 1

Exclusion Criteria:

* A history of life-threatening COPD including respiratory arrest, intensive care unit admission and/or requiring intubation.
* A history of more than one hospitalisation for COPD in the 2 years before Screening.
* Evidence of cor pulmonale, clinically significant pulmonary hypertension or chronic use of oxygen.
* Upper or lower respiratory tract infection, including exacerbation of COPD, requiring augmentation of therapy within 6 weeks of Screening.
* Other respiratory disorders: subjects with a history of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis or other chronic pulmonary diseases.
* A chest X-ray at Screening (or within 6 months prior to the Screening visit) showing abnormalities, which in the opinion of the Investigator are clinically significant and unrelated to COPD.
* A history of chronic disease including, but not limited to, unstable or uncontrolled hypertension (or been diagnosed with hypertension in the 6 months before Screening), sleep apnoea, cardiovascular, endocrine, neurological, hepatic, gastrointestinal, renal, haematological, urological, immunological or ophthalmic diseases that the Investigator believes are clinically significant e.g., unstable and could impact subject safety by participation in the study.
* Previous lung resection or lung reduction surgery.
* Vital sign assessments outside the following ranges: for inclusion blood pressure (after the subject is supine for 10 minutes) must be between 100 and 160 mmHg systolic, inclusive, and between 55 and 100 mmHg diastolic; heart rate must be between 40-100 bpm. These criteria must be met at Screening, Day -1 and pre-dose on Day 1.
* Have a clinical abnormality or laboratory parameters outside the reference range at Screening or Day -1.
* Liver function test results (ALT, aspartate amino transferase and gamma glutamyl transferase) >2 x ULN (upper limit of normal) at Screening or on Day -1.
* Chronic liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B virus (HBV) infection or hepatitis C antibodies.
* Unable or unwilling to undergo multiple venepuncture procedures or the subject has poor access to veins suitable for cannulation.
* If a woman, has a positive serum pregnancy test at Screening.
* Definite or suspected history of drug or alcohol abuse within the previous 5 years.
* Positive test for alcohol or drugs of abuse, including cannabinoids, alcohol, opiates, cocaine, amphetamines, benzodiazepines or barbiturates at Screening or on Day -1 or Day 1.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males, or >14 units for females.
* History of clinically significant allergies that, in the opinion of the Investigator would contraindicate their participation.
* Known allergy to the study drug or any of the excipients of the formulation or has previously been exposed to RV1729.
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study.
* Received an experimental drug or used an experimental medical device within 3 months or within a period less than five times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled.
* Requires routine treatment for COPD using one (or more) of the therapies listed in the protocol within the 6 weeks before Screening.
* A disclosed history or one known to the Investigator, of significant non-compliance in previous investigational studies or with prescribed medications.
* Has had major surgery, (requiring general anaesthesia) within 6 weeks before the Screening visit, or will not have fully recovered from surgery, or has planned surgery from Screening through to the end of the study. Note: subjects with planned surgical procedures to be conducted under local anaesthesia may participate.
* Employee of the Investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that Investigator or study centre, as well as family members of the employees or the Investigator.
* The subject is unable or unwilling to comply fully with the study protocol.
* The subject is mentally or legally incapacitated.
* Any other reason that the Investigator considers makes the subject unsuitable to participate.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 56 days
  Assessment of the number of adverse events reported by subjects following dosing
ECG assessment (12 lead ECG) | 56 days
  Change from pre-dose values
Vital sign assessment (blood pressure and heart rate) | 56 days
  Change from pre-dose values
Clinical laboratory assessments (blood and urine samples) | 56 days
  Change from pre-dose values
Spirometry assessment (FEV1 & FVC) | 56 days
  Change from pre-dose values
Use of rescue medication | 29 days
  Assessment of the number of occasions subjects are required to administer rescue medication
Peak expiratory flow (PEF) | 56 days
  Change from pre-dose values

SECONDARY OUTCOMES:
Plasma RV1729 levels | Days 1, 14 & 28 - 9 samples per day; Days 7, 21, 26 and 27 - 1 sample per day; Days 31 to 56 - 5 samples

OTHER OUTCOMES:
Serum biomarkers (measuring markers of inflammation in the blood) | Days 1, 14 & 28 - 3 samples per day; Days 7 & 21 - 1 sample per day; Day 56 - 1 sample
Exhaled breath condensate (measuring markers of oxidative stress) | Days 1, 14 & 28 - 2 samples per day
Sputum cell counts (measuring markers of inflammation in sputum) | Days 14, 21 & 26 - 1 sample per day
Pulmonary plethysmography (measuring airway resistance) | Days -1, 14 and 28 - 1 assessment per day

CONTACTS AND LOCATIONS:
Overall Officials: Liza O'Dowd, MD, Study Director — Sponsor GmbH
Locations (2):
- United Kingdom (2):
  - Belfast
  - Manchester